CLINICAL TRIAL: NCT02839070
Title: Influence of Sleep Regularity on Circadian Rhythms, Learning, Performance, and Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth Klerman MD PhD, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R01HL128538 (NIH)
Record Dates: First submitted 2016-07-15; First posted 2016-07-20 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Physiology
Keywords: Sleep; Learning; Circadian Rhythms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regular Schedule (Experimental): Participant will be on a regular sleep/wake schedule
  Interventions: Other: Sleep/Wake Schedule
- Irregular Schedule (Experimental): Participant will be on an irregular sleep/wake schedule
  Interventions: Other: Sleep/Wake Schedule

INTERVENTIONS:
Other: Sleep/Wake Schedule — Timing of sleep and wake

SUMMARY:
The study is a combination of outpatient and inpatient monitoring. During the 27-day inpatient portion of the study, the individual's sleep-wake schedule will be varied daily. Volunteers will be randomized to a regular or irregular inpatient schedule.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* BMI between 18.5 and 29.5

Exclusion Criteria:

* medications
* recent night-work, shift-work, or travel across >2 time zones
* use of medications
* pregnant or within 6 months post-partum

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2025-12 (Actual)

PRIMARY OUTCOMES:
Circadian phase | 27 days
  Circadian phase, as measured by melatonin, at end vs. beginning of inpatient portion of experiment
Learning | 27 days
  Sleep-dependent learning at 3-4 times during inpatient portion of the experiment
Mood | 27 days
  Mood (using a linear non-numeric scale) across difference days inpatient portion of the experiment

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth B Klerman, MD PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided